CLINICAL TRIAL: NCT04270760
Title: A Double-blind, Randomized, Placebo-controlled Phase 2 Study to Evaluate Efficacy, Safety, and Tolerability of Olpasiran (AMG 890) in Subjects With Elevated Lipoprotein(a)
Brief Title: Olpasiran Trials of Cardiovascular Events And LipoproteiN(a) Reduction - DOSE Finding Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20180109; 2019-003688-23 (EudraCT Number)
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Results first posted 2023-08-23 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Disease
Keywords: Olpasiran; AMG 890; siRNA; lipoprotein (a) Lp(a); Cardiovascular; Cardiovascular disease; Atherosclerotic cardiovascular disease; Cholesterol; Apolipoprotein (B); Hyperlipidemia; Dyslipidemia
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Hyperlipidemias; Dyslipidemias | interventions — olpasiran

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1 Olpasiran Dose 1 (Active Comparator)
  Interventions: Drug: Olpasiran
- Arm 2 Olpasiran Dose 2 (Active Comparator)
  Interventions: Drug: Olpasiran
- Arm 3 Olpasiran Dose 3 (Active Comparator)
  Interventions: Drug: Olpasiran
- Arm 4 Olpasiran Dose 4 (Active Comparator)
  Interventions: Drug: Olpasiran
- Arm 5 Placebo Dose 5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olpasiran — Dose 1 Dose 2 Dose 3 Dose 4
  Other Names: AMG 890
  Arms: Arm 1 Olpasiran Dose 1; Arm 2 Olpasiran Dose 2; Arm 3 Olpasiran Dose 3; Arm 4 Olpasiran Dose 4
Drug: Placebo — Dose 5
  Arms: Arm 5 Placebo Dose 5

SUMMARY:
Evaluate the effect of olpasiran administered subcutaneously (SC) compared with placebo, on percent change from baseline in lipoprotein(a) (Lp[a]).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years
* Lipoprotein (a) > 150 nmol/L
* Evidence of atherosclerotic cardiovascular disease

Exclusion Criteria:

* Severe renal dysfunction
* History or clinical evidence of hepatic dysfunction
* Malignancy within the last 5 years
* Currently receiving, or less than 3 months at Day 1 since receiving > 200 mg/day Niacin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2022-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (36):
- United States (12):
  - Westside Medical Associates of Los Angeles, Beverly Hills, California
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins, Baltimore, Maryland
  - New York University, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - Crossroads Clinical Research Inc, Mooresville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Protenium Clinical Research, Hurst, Texas
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Core Research Group Pty Ltd, Milton, Queensland
  - Monash Medical Centre, Clayton, Victoria
  - Linear Clinical Research Limited, Nedlands, Western Australia
  - Dr Heart Pty Ltd, Woolloongabba
- Canada (5):
  - LMC Clinical Research Incorporated, Brampton, Ontario
  - LMC Clinical Research Incorporated Thornhill, Concord, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Research Institute of McGill University Health Center - Glen Site, Montreal, Quebec
  - Clinique des Maladies Lipidiques de Quebec Incorporated, Québec, Quebec
- Denmark (3):
  - Aarhus Universitetshospital, Aarhus N
  - Herlev Gentofte Hospital, Herlev
  - Regionshospitalet Viborg, Viborg
- Thjonustumidstod Rannsoknaverkefna, Kopavogur, Iceland
- Japan (5):
  - Asahi General Hospital, Asahi-shi, Chiba
  - The Jikei University Kashiwa Hospital, Kashiwa-shi, Chiba
  - Asahikawa City Hospital, Asahikawa-shi, Hokkaido
  - Kanazawa Medical University Hospital, Kahoku-gun, Ishikawa-ken
  - Saitama Medical University Hospital, Iruma-gun, Saitama
- Netherlands (5):
  - Academisch Medisch Centrum, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Haga Ziekenhuis, The Hague
  - Universitair Medisch Centrum Utrecht, Utrecht
  - VieCuri Medisch Centrum, Venlo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] O'Donoghue ML, G Lopez JA, Knusel B, Gencer B, Wang H, Wu Y, Kassahun H, Sabatine MS. Study design and rationale for the Olpasiran trials of Cardiovascular Events And lipoproteiN(a) reduction-DOSE finding study (OCEAN(a)-DOSE). Am Heart J. 2022 Sep;251:61-69. doi: 10.1016/j.ahj.2022.05.004. Epub 2022 May 16. PMID 35588897
- [Background] O'Donoghue ML, Rosenson RS, Gencer B, Lopez JAG, Lepor NE, Baum SJ, Stout E, Gaudet D, Knusel B, Kuder JF, Ran X, Murphy SA, Wang H, Wu Y, Kassahun H, Sabatine MS; OCEAN(a)-DOSE Trial Investigators. Small Interfering RNA to Reduce Lipoprotein(a) in Cardiovascular Disease. N Engl J Med. 2022 Nov 17;387(20):1855-1864. doi: 10.1056/NEJMoa2211023. Epub 2022 Nov 6. PMID 36342163
- [Background] O'Donoghue ML, Rosenson RS, Lopez JAG, Lepor NE, Baum SJ, Stout E, Gaudet D, Knusel B, Kuder JF, Murphy SA, Wang H, Wu Y, Shah T, Wang J, Wilmanski T, Sohn W, Kassahun H, Sabatine MS; OCEAN(a)-DOSE Trial Investigators. The Off-Treatment Effects of Olpasiran on Lipoprotein(a) Lowering: OCEAN(a)-DOSE Extension Period Results. J Am Coll Cardiol. 2024 Aug 27;84(9):790-797. doi: 10.1016/j.jacc.2024.05.058. PMID 39168564
- [Background] Kaur G, Rosenson RS, Gencer B, Lopez JAG, Lepor NE, Baum SJ, Stout E, Gaudet D, Knusel B, Park JG, Wang H, Wu Y, Kassahun H, Sabatine MS, O'Donoghue ML. Olpasiran lowering of lipoprotein(a) according to baseline levels: insights from the OCEAN(a)-DOSE study. Eur Heart J. 2025 Mar 24;46(12):1162-1164. doi: 10.1093/eurheartj/ehae781. No abstract available. PMID 39565305
- [Background] Rosenson RS, Lopez JAG, Gaudet D, Baum SJ, Stout E, Lepor NE, Park JG, Murphy SA, Knusel B, Wang J, Wilmanski T, Wang H, Wu Y, Kassahun H, Sabatine MS, O'Donoghue ML; OCEAN(a)-DOSE Trial Investigators. Olpasiran, Oxidized Phospholipids, and Systemic Inflammatory Biomarkers: Results From the OCEAN(a)-DOSE Trial. JAMA Cardiol. 2025 May 1;10(5):482-486. doi: 10.1001/jamacardio.2024.5433. PMID 39937508
- [Derived] Karp A, Jacobs M, Barris B, Labkowsky A, Frishman WH. Lipoprotein(a): A Review of Risk Factors, Measurements, and Novel Treatment Modalities. Cardiol Rev. 2025 Jul-Aug 01;33(4):352-358. doi: 10.1097/CRD.0000000000000667. Epub 2024 Feb 28. PMID 38415744
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 34 centers in Australia, Denmark, Iceland, the Netherlands, Canada, the United States, and Japan between 28 July 2020 and 08 November 2022.
Pre-assignment Details: The Treatment Period was 48 weeks with investigational product (IP) administered subcutaneously (SC) every 12 weeks (Q12W) or 24 weeks (Q24W). After Week 48 there was an Extended Safety Follow-up Period without further dosing with IP for a minimum of 24 weeks. Participants remained on standard of care per their local guidelines during the Treatment Period and Extended Safety Follow-up Period.
Groups:
- Group 1: Olpasiran 10 mg Q12W: Participants were administered SC olpasiran 10 mg Q12W for 48 weeks with doses at Day 1, Week 12, Week 24, and Week 36. After Week 48 there was an Extended Safety Follow-up Period without further dosing with IP for a minimum of 24 weeks.
- Group 2: Olpasiran 75 mg Q12W: Participants were administered SC olpasiran 75 mg Q12W for 48 weeks with doses at Day 1, Week 12, Week 24, and Week 36. After Week 48 there was an Extended Safety Follow-up Period without further dosing with IP for a minimum of 24 weeks.
- Group 3: Olpasiran 225 mg Q12W: Participants were administered SC olpasiran 225 mg Q12W for 48 weeks with doses at Day 1, Week 12, Week 24, and Week 36. After Week 48 there was an Extended Safety Follow-up Period without further dosing with IP for a minimum of 24 weeks.
- Group 4: Olpasiran 225 mg Q24W: Participants were administered SC olpasiran 225 mg Q24W for 48 weeks with doses at Day 1 and Week 24. After Week 48 there was an Extended Safety Follow-up Period without further dosing with IP for a minimum of 24 weeks.
- Group 5: Placebo Q12W: Participants were administered SC placebo Q12W for 48 weeks with doses at Day 1, Week 12, Week 24, and Week 36. After Week 48 there was an Extended Safety Follow-up Period without further dosing with IP for a minimum of 24 weeks.
Period: Overall Study
Arm/Group | Group 1: Olpasiran 10 mg Q12W | Group 2: Olpasiran 75 mg Q12W | Group 3: Olpasiran 225 mg Q12W | Group 4: Olpasiran 225 mg Q24W | Group 5: Placebo Q12W
Started | 58 | 58 | 56 | 55 | 54
Entered Extended Safety Follow-up Period | 57 | 57 | 54 | 55 | 53
Completed | 57 | 55 | 52 | 55 | 53
Not Completed | 1 | 3 | 4 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): includes all randomized participants who received at least one dose of IP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Olpasiran 10 mg Q12W | Group 2: Olpasiran 75 mg Q12W | Group 3: Olpasiran 225 mg Q12W | Group 4: Olpasiran 225 mg Q24W | Group 5: Placebo Q12W | Total
Number analyzed (Participants) | 58 | 58 | 56 | 55 | 54 | 281
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.4 (9.5) | 61.3 (9.2) | 59.7 (10.1) | 61.8 (9.4) | 63.4 (8.9) | 61.9 (9.5)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 31 | 35 | 37 | 31 | 29 | 163
  65 - 74 years | 19 | 17 | 18 | 19 | 17 | 90
  75 - 84 years | 8 | 6 | 1 | 5 | 8 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 23 | 15 | 22 | 18 | 90
  Male | 46 | 35 | 41 | 33 | 36 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2 | 2 | 6
  Not Hispanic or Latino | 56 | 58 | 56 | 53 | 52 | 275
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 5 | 5 | 5 | 3 | 24
  Black or African American | 0 | 1 | 2 | 1 | 2 | 6
  White | 52 | 52 | 47 | 49 | 48 | 248
  Other | 0 | 0 | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Lipoprotein(a) (Lp[a]) at Week 36
Description: Least squares mean is from the repeated measures linear effects model which includes treatment group, stratification factors, scheduled visit and the interaction of treatment group with scheduled visit.
Time Frame: Baseline and Week 36
Population: Participants in the FAS with data available at each time point. FAS: includes all randomized participants who received at least one dose of IP.
Measure: Least Squares Mean (Standard Error); unit: Percentage Change in Lp(a)
Arm/Group | Group 1: Olpasiran 10 mg Q12W | Group 2: Olpasiran 75 mg Q12W | Group 3: Olpasiran 225 mg Q12W | Group 4: Olpasiran 225 mg Q24W | Group 5: Placebo Q12W
Number analyzed (Participants) | 57 | 57 | 53 | 53 | 51
Percentage Change in Lp(a) | -66.91 (1.78) | -93.78 (1.78) | -97.53 (1.82) | -96.89 (1.85) | 3.60 (1.89)
Statistical Analysis 1: Comparison: Group 1: Olpasiran 10 mg Q12W vs Group 5: Placebo Q12W; Group 1 versus (vs) Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model — Adjusted p-value is reported based on the Hochberg procedure to control the type I error for multiple comparisons. Each individual adjusted p-value is compared to 0.05 to determine statistical significance; Includes treatment group, stratification factors, scheduled visit and the interaction of treatment group with scheduled visit as covariates; Treatment difference = -70.51, 95% CI 2-sided [-75.12 to -65.90], Standard Error of Mean 2.35 — Treatment difference = percentage change in Group 1 - percentage change in Group 5 from Baseline at Week 36
Statistical Analysis 2: Comparison: Group 2: Olpasiran 75 mg Q12W vs Group 5: Placebo Q12W; Group 2 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Treatment difference = -97.38, 95% CI 2-sided [-101.98 to -92.77], Standard Error of Mean 2.35 — Treatment difference = percentage change in Group 2 - percentage change in Group 5 from Baseline at Week 36
Statistical Analysis 3: Comparison: Group 3: Olpasiran 225 mg Q12W vs Group 5: Placebo Q12W; Group 3 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Treatment difference = -101.13, 95% CI 2-sided [-105.79 to -96.47], Standard Error of Mean 2.38 — Treatment difference = percentage change in Group 3 - percentage change in Group 5 from Baseline at Week 36
Statistical Analysis 4: Comparison: Group 4: Olpasiran 225 mg Q24W vs Group 5: Placebo Q12W; Group 4 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -100.49, 95% CI 2-sided [-105.16 to -95.82], Standard Error of Mean 2.38 — Treatment difference = percentage change in Group 4 - percentage change in Group 5 from Baseline at Week 36

2. Secondary Outcome: Percentage Change From Baseline in Lp(a) at Week 48
Description: as for outcome 1
Time Frame: Baseline and Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage Change in Lp(a)
Arm/Group | Group 1: Olpasiran 10 mg Q12W | Group 2: Olpasiran 75 mg Q12W | Group 3: Olpasiran 225 mg Q12W | Group 4: Olpasiran 225 mg Q24W | Group 5: Placebo Q12W
Number analyzed (Participants) | 57 | 57 | 54 | 53 | 51
Percentage Change in Lp(a) | -64.89 (2.17) | -92.54 (2.17) | -97.29 (2.22) | -82.36 (2.25) | 3.59 (2.30)
Statistical Analysis 1: Comparison: Group 1: Olpasiran 10 mg Q12W vs Group 5: Placebo Q12W; Group 1 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -68.47, 95% CI 2-sided [-74.27 to -62.67], Standard Error of Mean 2.96 — Treatment difference = percentage change in Group 1 - percentage change in Group 5 from Baseline at Week 48
Statistical Analysis 2: Comparison: Group 2: Olpasiran 75 mg Q12W vs Group 5: Placebo Q12W; Group 2 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -96.12, 95% CI 2-sided [-101.92 to -90.33], Standard Error of Mean 2.96 — Treatment difference = percentage change in Group 2 - percentage change in Group 5 from Baseline at Week 48
Statistical Analysis 3: Comparison: Group 3: Olpasiran 225 mg Q12W vs Group 5: Placebo Q12W; Group 3 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -100.88, 95% CI 2-sided [-106.74 to -95.02], Standard Error of Mean 2.99 — Treatment difference = percentage change in Group 3 - percentage change in Group 5 from Baseline at Week 48
Statistical Analysis 4: Comparison: Group 4: Olpasiran 225 mg Q24W vs Group 5: Placebo Q12W; Group 4 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -85.94, 95% CI 2-sided [-91.83 to -80.06], Standard Error of Mean 3.00 — Treatment difference = percentage change in Group 4 - percentage change in Group 5 from Baseline at Week 48

3. Secondary Outcome: Percentage Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 36 and Week 48
Description: as for outcome 1
Time Frame: Baseline; Week 36 and Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage Change in LDL-C
Arm/Group | Group 1: Olpasiran 10 mg Q12W | Group 2: Olpasiran 75 mg Q12W | Group 3: Olpasiran 225 mg Q12W | Group 4: Olpasiran 225 mg Q24W | Group 5: Placebo Q12W
Number analyzed (Participants) | 57 | 57 | 54 | 53 | 51
Percentage Change in LDL-C
  Week 36: number analyzed (Participants) | 57 | 57 | 53 | 53 | 51
  Week 36 | -17.425 (4.258) | -16.284 (4.259) | -16.733 (4.389) | -18.462 (4.428) | 6.234 (4.520)
  Week 48: number analyzed (Participants) | 57 | 57 | 54 | 52 | 51
  Week 48 | -14.743 (4.419) | -11.481 (4.418) | -17.308 (4.532) | -16.908 (4.608) | 10.113 (4.688)
Statistical Analysis 1: Comparison: Group 1: Olpasiran 10 mg Q12W vs Group 5: Placebo Q12W; Week 36: Group 1 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -23.659, 95% CI 2-sided [-35.176 to -12.143], Standard Error of Mean 5.874 — Treatment difference = percentage change in Group 1 - percentage change in Group 5 from Baseline at Week 36
Statistical Analysis 2: Comparison: Group 2: Olpasiran 75 mg Q12W vs Group 5: Placebo Q12W; Week 36: Group 2 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -22.518, 95% CI 2-sided [-34.036 to -11.000], Standard Error of Mean 5.875 — Treatment difference = percentage change in Group 2 - percentage change in Group 5 from Baseline at Week 36
Statistical Analysis 3: Comparison: Group 3: Olpasiran 225 mg Q12W vs Group 5: Placebo Q12W; Week 36: Group 3 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -22.967, 95% CI 2-sided [-34.656 to -11.278], Standard Error of Mean 5.962 — Treatment difference = percentage change in Group 3 - percentage change in Group 5 from Baseline at Week 36
Statistical Analysis 4: Comparison: Group 4: Olpasiran 225 mg Q24W vs Group 5: Placebo Q12W; Week 36: Group 4 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -24.696, 95% CI 2-sided [-36.399 to -12.993], Standard Error of Mean 5.969 — Treatment difference = percentage change in Group 4 - percentage change in Group 5 from Baseline at Week 36
Statistical Analysis 5: Comparison: Group 1: Olpasiran 10 mg Q12W vs Group 5: Placebo Q12W; Week 48: Group 1 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -24.856, 95% CI 2-sided [-36.853 to -12.859], Standard Error of Mean 6.119 — Treatment difference = percentage change in Group 1 - percentage change in Group 5 from Baseline at Week 48
Statistical Analysis 6: Comparison: Group 2: Olpasiran 75 mg Q12W vs Group 5: Placebo Q12W; Week 48: Group 2 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -21.594, 95% CI 2-sided [-33.590 to -9.598], Standard Error of Mean 6.118 — Treatment difference = percentage change in Group 2 - percentage change in Group 5 from Baseline at Week 48
Statistical Analysis 7: Comparison: Group 3: Olpasiran 225 mg Q12W vs Group 5: Placebo Q12W; Week 48: Group 3 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -27.421, 95% CI 2-sided [-39.565 to -15.277], Standard Error of Mean 6.194 — Treatment difference = percentage change in Group 3 - percentage change in Group 5 from Baseline at Week 48
Statistical Analysis 8: Comparison: Group 4: Olpasiran 225 mg Q24W vs Group 5: Placebo Q12W; Week 48: Group 4 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -27.021, 95% CI 2-sided [-39.240 to -14.801], Standard Error of Mean 6.232 — Treatment difference = percentage change in Group 4 - percentage change in Group 5 from Baseline at Week 48

4. Secondary Outcome: Percentage Change From Baseline in Apolipoprotein (B) (ApoB) at Week 36 and Week 48
Description: as for outcome 1
Time Frame: Baseline; Week 36 and Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage Change in ApoB
Arm/Group | Group 1: Olpasiran 10 mg Q12W | Group 2: Olpasiran 75 mg Q12W | Group 3: Olpasiran 225 mg Q12W | Group 4: Olpasiran 225 mg Q24W | Group 5: Placebo Q12W
Number analyzed (Participants) | 57 | 57 | 54 | 53 | 52
Percentage Change in ApoB
  Week 36 | -11.496 (2.886) | -9.302 (2.885) | -10.241 (2.960) | -11.378 (3.012) | 7.394 (3.066)
  Week 48 | -7.748 (3.307) | -4.768 (3.305) | -7.218 (3.393) | -9.548 (3.443) | 12.292 (3.501)
Statistical Analysis 1: Comparison: Group 1: Olpasiran 10 mg Q12W vs Group 5: Placebo Q12W; Week 36: Group 1 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -18.890, 95% CI 2-sided [-26.303 to -11.477], Standard Error of Mean 3.779 — Treatment difference = percentage change in Group 1 - percentage change in Group 5 from Baseline at Week 36
Statistical Analysis 2: Comparison: Group 2: Olpasiran 75 mg Q12W vs Group 5: Placebo Q12W; Week 36: Group 2 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -16.696, 95% CI 2-sided [-24.107 to -9.284], Standard Error of Mean 3.778 — Treatment difference = percentage change in Group 2 - percentage change in Group 5 from Baseline at Week 36
Statistical Analysis 3: Comparison: Group 3: Olpasiran 225 mg Q12W vs Group 5: Placebo Q12W; Week 36: Group 3 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -17.635, 95% CI 2-sided [-25.139 to -10.131], Standard Error of Mean 3.825 — Treatment difference = percentage change in Group 3 - percentage change in Group 5 from Baseline at Week 36
Statistical Analysis 4: Comparison: Group 4: Olpasiran 225 mg Q24W vs Group 5: Placebo Q12W; Week 36: Group 4 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -18.772, 95% CI 2-sided [-26.303 to -11.241], Standard Error of Mean 3.839 — Treatment difference = percentage change in Group 4 - percentage change in Group 5 from Baseline at Week 36
Statistical Analysis 5: Comparison: Group 1: Olpasiran 10 mg Q12W vs Group 5: Placebo Q12W; Week 48: Group 1 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -20.040, 95% CI 2-sided [-28.757 to -11.323], Standard Error of Mean 4.443 — Treatment difference = percentage change in Group 1 - percentage change in Group 5 from Baseline at Week 48
Statistical Analysis 6: Comparison: Group 2: Olpasiran 75 mg Q12W vs Group 5: Placebo Q12W; Week 48: Group 2 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -17.060, 95% CI 2-sided [-25.774 to -8.345], Standard Error of Mean 4.442 — Treatment difference = percentage change in Group 2 - percentage change in Group 5 from Baseline at Week 48
Statistical Analysis 7: Comparison: Group 3: Olpasiran 225 mg Q12W vs Group 5: Placebo Q12W; Week 48: Group 3 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -19.509, 95% CI 2-sided [-28.336 to -10.682], Standard Error of Mean 4.500 — Treatment difference = percentage change in Group 3 - percentage change in Group 5 from Baseline at Week 48
Statistical Analysis 8: Comparison: Group 4: Olpasiran 225 mg Q24W vs Group 5: Placebo Q12W; Week 48: Group 4 vs Group 5; Test type: Superiority; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 1, analysis 1]; Treatment difference = -21.839, 95% CI 2-sided [-30.700 to -12.979], Standard Error of Mean 4.517 — Treatment difference = percentage change in Group 4 - percentage change in Group 5 from Baseline at Week 48

5. Secondary Outcome: Mean Serum Olpasiran Concentrations at Day 1, Week 24 and Week 48
Description: Pharmacokinetic blood draws were collected at one timepoint during the 6-12 and 24-72 hour flexible time windows and at Week 48.
  Lower limit of quantification (LLOQ) = 0.400 ng/mL. Values below the LLOQ were set to zero.
Time Frame: Pre-dose and 1, 3, 6-12, and 24-72 hours post-dose on Day 1 and Week 24; Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1: Olpasiran 10 mg Q12W | Group 2: Olpasiran 75 mg Q12W | Group 3: Olpasiran 225 mg Q12W | Group 4: Olpasiran 225 mg Q24W
Number analyzed (Participants) | 55 | 56 | 49 | 52
ng/mL
  Day 1: Pre-dose: number analyzed (Participants) | 54 | 52 | 47 | 51
  Day 1: Pre-dose | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 1: 1 Hour Post-dose: number analyzed (Participants) | 52 | 44 | 45 | 46
  Day 1: 1 Hour Post-dose | 12.3 (6.9) | 67.1 (47.4) | 220 (218) | 275 (450)
  Day 1: 3 Hours Post-dose: number analyzed (Participants) | 53 | 44 | 44 | 48
  Day 1: 3 Hours Post-dose | 18 (9.85) | 80.3 (43.2) | 291 (273) | 324 (383)
  Day 1: 6-12 Hours Post-dose: number analyzed (Participants) | 8 | 9 | 8 | 16
  Day 1: 6-12 Hours Post-dose | 18.6 (10.1) | 61.7 (36) | 420 (432) | 329 (191)
  Day 1: 24-72 Hours Post-dose: number analyzed (Participants) | 11 | 12 | 9 | 17
  Day 1: 24-72 Hours Post-dose | 0.995 (0.946) | 20.4 (13.2) | 63.2 (59.7) | 103 (47.3)
  Week 24: Pre-dose | 0.00 (0.00) | 0.0315 (0.134) | 0.498 (1.88) | 0.0645 (0.22)
  Week 24: 1 Hour Post-dose: number analyzed (Participants) | 52 | 48 | 48 | 45
  Week 24: 1 Hour Post-dose | 12.4 (7.23) | 73.6 (43.6) | 204 (144) | 253 (247)
  Week 24: 3 Hours Post-dose: number analyzed (Participants) | 53 | 49 | 46 | 48
  Week 24: 3 Hours Post-dose | 16.3 (9.2) | 96.3 (63.5) | 278 (193) | 332 (255)
  Week 24: 6-12 Hours Post-dose: number analyzed (Participants) | 8 | 10 | 7 | 15
  Week 24: 6-12 Hours Post-dose | 17.2 (10.2) | 76.3 (54.7) | 271 (229) | 315 (191)
  Week 24: 24-72 Hours Post-dose: number analyzed (Participants) | 7 | 9 | 8 | 16
  Week 24: 24-72 Hours Post-dose | 1.27 (1.82) | 17.3 (18.9) | 99 (59.1) | 96.3 (50.3)
  Week 48: number analyzed (Participants) | 52 | 50 | 48 | 51
  Week 48 | 0.00 (0.00) | 0.0599 (0.168) | 0.533 (0.592) | 0.127 (0.693)

ADVERSE EVENTS:
Time Frame: Treatment Period: Median duration was 11.07 months. Extended Safety Follow-up Period: Median duration was 8.56 months.
Description: FAS: includes all randomized participants who received at least one dose of IP. For safety analysis FAS was used based on actual treatment received.
Groups:
- Group 1; Treatment Period: Olpasiran 10 mg Q12W: Participants were administered SC olpasiran 10 mg Q12W for 48 weeks with doses at Day 1, Week 12, Week 24, and Week 36.
- Group 2; Treatment Period: Olpasiran 75 mg Q12W: Participants were administered SC olpasiran 75 mg Q12W for 48 weeks with doses at Day 1, Week 12, Week 24, and Week 36.
- Group 3; Treatment Period: Olpasiran 225 mg Q12W: Participants were administered SC olpasiran 225 mg Q12W for 48 weeks with doses at Day 1, Week 12, Week 24, and Week 36.
- Group 4; Treatment Period: Olpasiran 225 mg Q24W: Participants were administered SC olpasiran 225 mg Q24W for 48 weeks with doses at Day 1 and Week 24.
- Group 5; Treatment Period: Placebo Q12W: Participants were administered SC placebo Q12W for 48 weeks with doses at Day 1, Week 12, Week 24, and Week 36.
- Group 1; Extended Safety Follow-up Period: Olpasiran 10 mg Q12W; Group 2; Extended Safety Follow-up Period: Olpasiran 75 mg Q12W; Group 3; Extended Safety Follow-up Period: Olpasiran 225 mg Q12W; Group 4; Extended Safety Follow-up Period: Olpasiran 225 mg Q24W; Group 5; Extended Safety Follow-up: Placebo Q12W: After Week 48 there was an extended safety follow-up without further dosing with IP for a minimum of 24 weeks.
Arm/Group | Group 1; Treatment Period: Olpasiran 10 mg Q12W | Group 2; Treatment Period: Olpasiran 75 mg Q12W | Group 3; Treatment Period: Olpasiran 225 mg Q12W | Group 4; Treatment Period: Olpasiran 225 mg Q24W | Group 5; Treatment Period: Placebo Q12W | Group 1; Extended Safety Follow-up Period: Olpasiran 10 mg Q12W | Group 2; Extended Safety Follow-up Period: Olpasiran 75 mg Q12W | Group 3; Extended Safety Follow-up Period: Olpasiran 225 mg Q12W | Group 4; Extended Safety Follow-up Period: Olpasiran 225 mg Q24W | Group 5; Extended Safety Follow-up: Placebo Q12W
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58 | 0/56 | 0/55 | 1/54 | 0/57 | 0/57 | 0/54 | 0/55 | 0/53
Serious Adverse Events (participants affected / at risk) | 3/58 | 3/58 | 6/56 | 4/55 | 8/54 | 4/57 | 2/57 | 6/54 | 5/55 | 4/53
Other Adverse Events (participants affected / at risk) | 35/58 | 40/58 | 37/56 | 36/55 | 29/54 | 18/57 | 25/57 | 21/54 | 17/55 | 17/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1; Treatment Period: Olpasiran 10 mg Q12W (N=58) | Group 2; Treatment Period: Olpasiran 75 mg Q12W (N=58) | Group 3; Treatment Period: Olpasiran 225 mg Q12W (N=56) | Group 4; Treatment Period: Olpasiran 225 mg Q24W (N=55) | Group 5; Treatment Period: Placebo Q12W (N=54) | Group 1; Extended Safety Follow-up Period: Olpasiran 10 mg Q12W (N=57) | Group 2; Extended Safety Follow-up Period: Olpasiran 75 mg Q12W (N=57) | Group 3; Extended Safety Follow-up Period: Olpasiran 225 mg Q12W (N=54) | Group 4; Extended Safety Follow-up Period: Olpasiran 225 mg Q24W (N=55) | Group 5; Extended Safety Follow-up: Placebo Q12W (N=53)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site urticaria (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis intestinal perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant melanoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device inappropriate shock delivery (Product Issues) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinoma (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1; Treatment Period: Olpasiran 10 mg Q12W (N=58) | Group 2; Treatment Period: Olpasiran 75 mg Q12W (N=58) | Group 3; Treatment Period: Olpasiran 225 mg Q12W (N=56) | Group 4; Treatment Period: Olpasiran 225 mg Q24W (N=55) | Group 5; Treatment Period: Placebo Q12W (N=54) | Group 1; Extended Safety Follow-up Period: Olpasiran 10 mg Q12W (N=57) | Group 2; Extended Safety Follow-up Period: Olpasiran 75 mg Q12W (N=57) | Group 3; Extended Safety Follow-up Period: Olpasiran 225 mg Q12W (N=54) | Group 4; Extended Safety Follow-up Period: Olpasiran 225 mg Q24W (N=55) | Group 5; Extended Safety Follow-up: Placebo Q12W (N=53)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 2 | 2 | 1 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 3 | 1 | 4 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 3
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 3 | 1 | 0 | 0 | 0 | 2 | 1
Fatigue (General disorders) | 6 | 8 | 3 | 2 | 3 | 2 | 1 | 0 | 0 | 1
Injection site bruising (General disorders) | 0 | 4 | 5 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 3 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 2 | 3 | 1 | 5 | 2 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 2 | 1 | 4 | 1 | 2 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 1 | 1 | 3 | 0 | 0 | 1 | 2 | 0 | 0
Immunisation reaction (Immune system disorders) | 8 | 4 | 2 | 4 | 5 | 0 | 0 | 2 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 8 | 7 | 4 | 6 | 8 | 11 | 14 | 10 | 10
Gastroenteritis (Infections and infestations) | 1 | 4 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2 | 4 | 1 | 1 | 3 | 1 | 0 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 3 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 2 | 1 | 2 | 2 | 2 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 4 | 2 | 1 | 1 | 0 | 4 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 3 | 1 | 2 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 3 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 3 | 1 | 2 | 2 | 1 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3 | 2 | 1 | 0 | 1 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 5 | 7 | 1 | 3 | 3 | 1 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4 | 4 | 4 | 2 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 0
Areflexia (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 2 | 1 | 2 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 6 | 7 | 6 | 6 | 4 | 0 | 1 | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3
Hypertension (Vascular disorders) | 4 | 2 | 3 | 2 | 2 | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT04270760/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT04270760/SAP_001.pdf